CLINICAL TRIAL: NCT03676842
Title: Prospective Study for the Treatment of Atherosclerotic Lesions in the Superficial Femoral And/or Popliteal Arteries Using the FLEX Scoring Catheter Plus DCB
Acronym: FORTEZ
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment- Hospital during COVID
Sponsor: VentureMed Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The FORTEZ Study
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- FLEX Scoring Catheter plus DCB (Experimental): This is a single-arm study. All patients will be treated with the FLEX Scoring Catheter followed by an IN.PACT Admiral Drug-Coated Balloon (Medtronic Vascular; Galway, Ireland).
  Interventions: Combination Product: FLEX Dynamic Scoring Catheter with IN.PACT Admiral DCB

INTERVENTIONS:
Combination Product: FLEX Dynamic Scoring Catheter with IN.PACT Admiral DCB — Treatment by the FLEX Scoring Catheter followed by an IN.PACT Admiral DCB

SUMMARY:
Prospective, single-center, single-arm, non-randomized study to assess the safety and efficacy of the FLEX Scoring Catheter in patients with atherosclerotic peripheral artery disease in the superficial femoral and popliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

* Women of child-bearing potential must have a negative test within 7 days of the initial procedure
* Patient or patient's legal representative has been informed of the nature of the study, agrees to participate and comply with all follow-up visits, and has signed the informed consent.
* Patient is eligible for standard surgical repair in the target limb if necessary.
* Patient has Rutherford Clinical Category estimated as 2-6.
* A life expectancy >1 year.

Angiographic Inclusion Criteria:

* Target lesion(s) is located within the SFA and/or the popliteal arteries.
* Target lesion has >70% stenosis by visual assessment.
* The reference vessel diameter is between 4-6 mm.
* One long or multiple serial lesions.
* de novo or non-stented re-stenotic lesions.
* At least one BTK artery patent to the ankle.
* Successful treatment of iliac inflow stenosis to the target limb. Stenosis can be treated during the same procedure using standard angioplasty and/or stenting but atherectomy is excluded. The inflow lesion(s) must be treated first, before consideration of treatment of the target lesion. Subject can be enrolled if the treated inflow lesion(s) results in <30% residual stenosis and no evidence of embolization or significant complications.

Exclusion Criteria:

* Rutherford Clinical Category 1.
* Previously implanted ipsilateral femoral or popliteal stent.
* Evidence of aneurysm or acute thrombus in the target vessel.
* Patients with previous bypass surgery in the lower target extremity.
* Planned major amputation, above the ankle, of either limb.
* Patient has significant stenosis or occlusion of inflow tract not successfully treated (>30% residual stenosis and/or significant complication of the procedure)
* History of any open surgical procedure within the past 30 days
* Planned endovascular or vascular surgery procedure within 14 days prior to the ATK procedure, except to treat the inflow vessels on the day of the procedure, or within the next 30 days after the ATK procedure on the target limb.
* Patient has an allergy to contrast medium that cannot be adequately pretreated.
* Episode of acute limb ischemia within the past 30 days.
* Patient has systemic infection with positive blood cultures/bacteremia within one week
* Patient has hypercoagulable disorder.
* Patient is contraindicated for antiplatelet, anticoagulant, or thrombolytic therapy.
* Myocardial infarction within 30 days prior to enrollment.
* History of stroke or TIA within 90 days prior to enrollment.
* Patient has acute or chronic renal disease (i.e., as measured by a serum creatinine of >2.5 mg/dL or >220 umol/L)
* Patient is pregnant or breastfeeding
* Patient is participating in another research study of a device, medication, which could, in the opinion of the investigator, affect the results of this study.
* Patient has other medical, social, or psychological problems that in the opinion of the investigator, would preclude them from receiving this treatment and the procedure and or participating in evaluations pre- and post-treatment.
* Thrombolysis of the target lesion within 72 hours prior to the initial procedure, where complete resolution of the thrombus was not achieved.
* Known allergies to both antiplatelet, aspirin, or heparin.
* History of neutropenia, coagulopathy, or thrombocytopenia that was unexplained or is considered to be a risk for reoccurrence.
* Platelet count less than 80,000/uL
* Patient requires general anesthesia for procedure.
* Patient requires dialysis.

Angiographic Exclusion Criteria:

* Acute Total Occlusions; evidence of acute thrombus formation by angiography.
* Severe calcification of target lesion described as circumferential calcium and >50% of lesion length.
* Sub-intimal access required.
* Inability to cross the lesion with a guidewire.
* Atherectomy in the target lesion, target artery or for inflow treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Technical feasibility of the FLEX Scoring Catheter | Through study completion: Approximately 12 months
  Evaluation of the technical feasibility of using the FLEX Scoring Catheter during the endovascular treatment of critical SFA or popliteal artery lesions.

SECONDARY OUTCOMES:
Absence of lesion restenosis | 6 and 12 months
  Defined by PSVR ≥ to 2.5 at duplex scan
Change in Rutherford Class of symptom | 6 and 12 months
Change in ankle-brachial index (ABI) | 6 and 12 months
Absence of clinically driven target vessel revascularization | 12 months
Major adverse events (MAE) | at procedure, 6 months, and 12 months
Proportion of luminal gain | at procedure
Proportion of stent implantation | at procedure
Proportions and classifications of dissections | at procedure

CONTACTS AND LOCATIONS:
Overall Officials: Louis Lopez, MD, Principal Investigator — Allen County Cardiology
Locations (1):
- Saint Joseph Hospital, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No